CLINICAL TRIAL: NCT07282457
Title: A Prospective, Randomized, Sham-controlled, Dose-finding Phase 1/2 Two-part Trial to Evaluate the Safety, Tolerability, and Efficacy of ZM-02 Injection in Patients With Advanced Retinitis Pigmentosa
Brief Title: Prospective, Randomized, Sham-controlled, Dose-finding I/II Trial of Safety and Efficacy of Modified Optogenetic Gene Therapy (ZM-02 Injection)
Acronym: PRISM
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhongmou Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZM-02-201
Record Dates: First submitted 2025-11-26; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Retinitis Pigmentosa (RP)
Keywords: gene therapy; AAV; RP; optogenetics
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose ZM-02 (Experimental)
  Interventions: Genetic: ZM-02 (low dose)
- High Dose ZM-02 (Experimental)
  Interventions: Genetic: ZM-02 (high dose)
- ZM-02 (selected dose) (Experimental)
  Interventions: Genetic: ZM-02 (selected dose)
- Sham Comparator (Sham Comparator)
  Interventions: Procedure: Sham injection

INTERVENTIONS:
Genetic: ZM-02 (low dose) — Single unilateral IVT injection of low-dose ZM-02 in the study eye
  Arms: Low Dose ZM-02
Genetic: ZM-02 (high dose) — Single unilateral IVT injection of high-dose ZM-02 in the study eye
  Arms: High Dose ZM-02
Genetic: ZM-02 (selected dose) — Single unilateral IVT injection of selected-dose ZM-02 in the study eye
  Arms: ZM-02 (selected dose)
Procedure: Sham injection — Sham IVT procedure in the study eye
  Arms: Sham Comparator

SUMMARY:
This is a Phase 1/2, multi-center, randomized, sham-controlled, dose-escalation study evaluating ZM-02 in patients with advanced retinitis pigmentosa (RP).

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is the most common inherited retinal disease, characterized by progressive loss of visual function that can lead to severe visual impairment or blindness with no effective treatment.

This Phase 1/2 study is designed to evaluate the safety, tolerability, and preliminary efficacy of a single unilateral intravitreal injection of ZM-02 at escalating dose levels in patients with advanced RP. The study includes a sham-controlled design and will assess safety outcomes as well as multiple functional and structural measures of visual performance over long-term follow-up.

ELIGIBILITY:
Inclusion Criteria

1. Male or female participants aged 6 to 60 years.
2. Clinical diagnosis of advanced retinitis pigmentosa (RP).
3. Best corrected visual acuity at or below the protocol-defined threshold in the study eye.
4. Presence of sufficient retinal structure in the study eye as determined by screening assessments.
5. Ability to understand and sign informed consent (and assent, when applicable).

Exclusion Criteria

1. Presence of other ocular conditions that could interfere with study assessments.
2. History of significant ocular surgery in the study eye within a protocol-defined period.
3. Active ocular infection or inflammation.
4. Clinically significant systemic disease that could increase study risk or interfere with assessments.
5. Positive screening for clinically significant infectious diseases, as defined in the protocol.
6. Pregnant or breastfeeding individuals.
7. Any condition that, in the investigator's judgment, would make the participant unsuitable for study participation.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2029-12-25 (Estimated); Study Completion 2031-12-25 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of ZM-02 | Baseline to Week 52.
  Incidence of severity of ocular and systemic adverse events (AEs) and serious adverse events (SAEs) following a single intravitreal injection of ZM-02.

SECONDARY OUTCOMES:
Change from Baseline in Best-Corrected Visual Acuity (BCVA) of Both Eyes | Baseline to Week 52.
Change from Baseline in Functional Vision (MLMT) | Baseline to Week 52.
  Change from baseline in the multi-luminance mobility test (MLMT) performance.
Change from Baseline in Vision-Related Quality of Life (NEI VFQ-25) | Baseline to Week 52.

IPD SHARING:
Plan to Share IPD: No